CLINICAL TRIAL: NCT02947854
Title: An Open-label, Phase I/Proof of Principle, Dose Escalation Study to Assess Safety, Tolerability and Immune Response of Fimaporfin-induced Photochemical Internalisation (PCI) of Antigen/Adjuvant in Healthy Male/Female Subjects
Brief Title: Study to Assess Safety, Tolerability and Immune Response of Fimaporfin-induced Photochemical Internalisation of Antigen/Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCIA102-16
Record Dates: First submitted 2016-10-12; First posted 2016-10-28 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteer
Keywords: Vaccine; Photochemical Internalisation; Immune Response; Peptide vaccine; Anti cancer vaccine
MeSH Terms: interventions — Photosensitizing Agents; poly ICLC; Peptides; keyhole-limpet hemocyanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Photosensitizer and adjuvant (Experimental): Run-in cohort for selection of fimaporfin starting dose in the main study. Single intradermal dosing of fimaporfin and adjuvant (Hiltonol [poly-ICLC]) followed by light application.
  Interventions: Drug: Fimaporfin (Photosensitizer); Biological: Hiltonol (Poly-ICLC)
- Photosensitizer, adjuvant and antigens (Experimental): Main part: Intradermal dosing of fimaporfin, adjuvant (Hiltonol, poly-ICLC) and antigens (KLH and HPV E7) followed by light application.
  Interventions: Drug: Fimaporfin (Photosensitizer); Biological: Hiltonol (Poly-ICLC); Biological: HPV E7 (Human Papilloma Virus E7) peptides; Biological: KLH (Keyhole Limpet Hemocyanin)
- Assessments of time between ID dosing and light (Experimental): Optional part: Assessment of different time interval between intradermal dosing of fimaporfin, adjuvant/antigens and light application.
  Interventions: Drug: Fimaporfin (Photosensitizer); Biological: Hiltonol (Poly-ICLC); Biological: HPV E7 (Human Papilloma Virus E7) peptides; Biological: KLH (Keyhole Limpet Hemocyanin)

INTERVENTIONS:
Drug: Fimaporfin (Photosensitizer)
Biological: Hiltonol (Poly-ICLC)
Biological: HPV E7 (Human Papilloma Virus E7) peptides
  Arms: Assessments of time between ID dosing and light; Photosensitizer, adjuvant and antigens
Biological: KLH (Keyhole Limpet Hemocyanin)
  Arms: Assessments of time between ID dosing and light; Photosensitizer, adjuvant and antigens

SUMMARY:
Fimaporfin (TPCS2a) is a photosensitiser drug being developed by PCI Biotech AS for use in novel Photochemical Internalisation (PCI) technology. PCI technology is designed to enhance the effects of other drugs in a site-specific, light-directed manner and is used to re-localise endocytosed molecules from endosomes to cytosol. This research study is evaluating the use of the PCI Technology in combination with adjuvant and vaccine antigens for safety and induction of immune responses.

ELIGIBILITY:
Inclusion Criteria

1. Subjects will be; 1.1. males or females 1.2. Caucasian 1.3. between 18 and 55 years of age, inclusive
2. Subjects will have a 2.1. body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive 2.2. body weight between 50 and 100 kg, inclusive
3. Subjects will be in good health, as determined by; 3.1. medical history, 3.2. physical examination, 3.3. vital signs assessment, 3.4. 12-lead electrocardiogram (ECG) 3.5. clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinaemia is acceptable)
4. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria

1. Male subjects who do not agree, or whose partners of childbearing potential do not agree, to use appropriate contraception (ie, a condom with spermicidal foam/gel/film/cream/suppository) or to refrain from donating sperm from the time of the first dose until 3 months after the final dose administration.

   1.1. Male subjects whose partners of childbearing potential do not agree to use an additional acceptable method of contraception.
2. Female subjects of childbearing potential who do not agree to use 2 acceptable methods of contraception from the time of screening until 3 months after the final dose administration.
3. Subjects who have a negative result for the test for human leukocyte antigen (HLA)-A2 (Parts B and C only).
4. Subjects who have donated; 4.1. blood in the 3 months prior to screening, 4.2. plasma in the 7 days prior to screening, 4.3. platelets in the 6 weeks prior to screening.
5. Subjects who; 5.1. consume more than 28 units of alcohol per week if male 5.2. consume more than 21 units of alcohol per week if female 5.3. have a significant history of alcoholism or drug/chemical abuse, as determined by the Investigator Note: 1 unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine or 25 mL of spirits
6. Subjects who smoke more than 10 cigarettes or use the equivalent in tobacco per day.
7. Subjects who have used the following within 7 days of first dose (use of intermittent paracetamol ≤2 g/day is acceptable), unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety:

   7.1. any non-prescribed systemic or topical medication 7.2. any herbal remedy 7.3. any vitamin supplement 7.4. any mineral supplement
8. Subjects who have received; 8.1. any prescribed systemic or topical medication (including steroids) within 14 days of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.

   8.2. slow-release medicinal formulations considered to still be active within 14 days of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
9. Subjects who have received a vaccine within 3 months of first dose administration.
10. Subjects who have an abnormality in heart rate, blood pressure, temperature, or respiration rate at screening and prior to first dose that in the opinion of the Investigator increases the risk of participating in the study.
11. Subjects who have; 11.1. a positive urine drugs of abuse screen (confirmed by repeat) at screening or first admission.

    11.2. a positive alcohol breath test (confirmed by repeat) at screening or first admission.
12. Subjects who have an abnormality in the 12-lead ECG at screening and prior to first dose that in the opinion of the Investigator increases the risk of participating in the study.
13. Subjects who are pregnant, breastfeeding, or lactating.
14. Subjects who are still participating in another clinical study (eg, attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to first dose administration.
15. Subjects who have previously been exposed to KLH antigen (Parts B and C only).
16. Subjects who have a known previous exposure to HVP E7 (Parts B and C only).
17. Subjects who have a significant history of drug allergy, as determined by the Investigator.
18. Subjects who have a known allergy or sensitivity to Hiltonol and/or photosensitisers.
19. Subjects who have any clinically significant abnormal physical examination finding, as determined by the Investigator.
20. Subjects who have any clinically significant medical history, as determined by the Investigator.
21. Subjects who have any clinically significant allergic condition (excluding non-active hayfever), as determined by the Investigator.
22. Subjects with porphyria or hypersensitivity to porphyrins.
23. Subjects who have, or who have a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, immunological or other major disorder, as determined by the Investigator.
24. Subjects who have had a clinically significant illness within 4 weeks of first dose, as determined by the Investigator.
25. Subjects who have any clinically significant abnormal laboratory safety findings at screening and prior to first dose, as determined by the Investigator (1 repeat assessment is acceptable at each timepoint).
26. Subjects who have a C-reactive protein value that is above the upper limit of normal at screening and prior to first dose (1 repeat assessment is acceptable at each timepoint).
27. Subjects who; 27.1. have serum hepatitis, 27.2. are carriers of the hepatitis B surface antigen (HBsAg), 27.3. are carriers of the hepatitis C antibody, 27.4. have a positive result for the test for human immunodeficiency virus (HIV) antibodies.
28. Subjects who have tattoos, scars, or moles that in the opinion of the Investigator are likely to interfere with dosing or study assessments at any of the potential dosing sites (upper arms or abdomen).
29. Subjects who have previously taken part in or withdrawn from this study.
30. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Up to 1 year
  Safety
Incidence of abnormal and clinical significant measures | Up to 1 year
  Clinical Laboratory, ECG, Vital Signs and Physical Examinations
Pain as measured by Visual Analogue Scale (VAS) | Up to 1 year
  Tolerability
Incidence and grading of local skin reactions as by CTCAE v. 4.03 | Up to 1 year
  Local Tolerability (pain, erythema, oedema, induration and ulceration)

SECONDARY OUTCOMES:
Induction of Immune Response | Up to 1 year
  Blood samples will be collected prior, during and after treatment for assessment of Antibody Production and T-cell Responses (change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, MRCS, MFPM, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit Limited, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otterhaug T, Janetzki S, Welters MJP, Hakerud M, Nedberg AG, Edwards VT, Boekestijn S, Loof NM, Selbo PK, Olivecrona H, van der Burg SH, Hogset A. Photochemical Internalization Enhanced Vaccination Is Safe, and Gives Promising Cellular Immune Responses to an HPV Peptide-Based Vaccine in a Phase I Clinical Study in Healthy Volunteers. Front Immunol. 2021 Jan 8;11:576756. doi: 10.3389/fimmu.2020.576756. eCollection 2020. PMID 33488576
- See also: Sponsor — http://pcibiotech.no/